CLINICAL TRIAL: NCT04204096
Title: A Phase III, Multicenter, Observer Blind, Randomized, Controlled Study to Evaluate Immune Equivalence of Multi-dose Formulation Against Single-dose Formulation of Vi-DT Typhoid Conjugate Vaccine and Safety in Healthy Filipino......
Brief Title: Immune Equivalence Between Multi-dose and Single Dose Formulation of Vi-DT and Their Overall Safety (Phase III)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: International Vaccine Institute (Other)
Collaborators: SK Bioscience Co., Ltd. (Industry); Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IVI T004
Record Dates: First submitted 2019-12-17; First posted 2019-12-18 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Typhoid
Keywords: Typhoid conjugate vaccine; Vi-DT; Safety; Immunogenicity
MeSH Terms: conditions — Typhoid Fever | interventions — Diphtheria Toxoid; Dosage Forms

STUDY DESIGN:
Intervention Model Description: Participants age 6 months to 45 years
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study is observer blind:
  1. Vaccine administrator and vaccine safety evaluator at site will be two distinct persons.
  2. Laboratory personnel who analyzes immunogenicity at sponsor is also blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vi-DT Multi-dose (Experimental): * 750 participants (6 mo - 45 yrs)
  * Dose: 0.5mL, Vi polysaccharide typhoid vaccine conjugated with Diphtheria toxoid protein (Vi-DT), manufactured by SK bioscience (Republic of Korea)
  * Dosage form: Liquid, 25µg Vi polysaccharide/0.5mL, presented in Type I glass vial (multi-dose formulation Vi-DT contains preservative 2 PE)
  * Mode of Administration: Intramuscular injection
  * Frequency of administration: Once
  Interventions: Biological: Vi-DT (Multi-dose formulation)
- Vi-DT Single-dose (Experimental): * 750 participants (6 mo - 45 yrs)
  * Dose: 0.5mL, Vi polysaccharide typhoid vaccine conjugated with Diphtheria toxoid protein (Vi-DT), manufactured by SK bioscience (Republic of Korea)
  * Dosage form: Liquid, 25µg Vi polysaccharide/0.5mL, presented in Type I glass vial (single dose formulation Vi-DT without any preservative)
  * Mode of Administration: Intramuscular injection
  * Frequency of administration: Once
  Interventions: Biological: Vi-DT (Single dose formulation)
- Control (Active Comparator): * 300 participants (6 mo - 45 yrs)
  * Dose: 0.5mL, Locally available Meningococcal conjugate vaccine
  * Dosage form: Lyophilized white powder
  * Mode of Administration: Intramuscular injection
  * Frequency of administration: Once (For participants 6 months to 1 year, one more dose will be provided after the study unblinding)
  Interventions: Biological: Control Vaccine

INTERVENTIONS:
Biological: Vi-DT (Multi-dose formulation) — * Manufacturer: SK bioscience Co., Ltd.
  * Dose formulation: 25 µg Vi polysaccharide /0.5 mL, presented in Type I glass vial (multi dose Vi-DT with preservative 2 PE)
  * Mode of Administration: 0.5 mL by intramuscular injection in the left anterolateral thigh or left arm deltoid region in participants below 2 years of age, less dominant arm deltoid region in age group 2 to 45 years
  * Storage Conditions: +2 to +8°C
  Other Names: Vi polysaccharide typhoid vaccine conjugated with Diphtheria toxoid protein
  Arms: Vi-DT Multi-dose
Biological: Vi-DT (Single dose formulation) — * Manufacturer: SK bioscience Co., Ltd.
  * Dose formulation: 25 µg Vi polysaccharide /0.5 mL, presented in Type I glass vial (single dose Vi-DT without any preservative)
  * Mode of Administration: 0.5 mL by intramuscular injection in the left anterolateral thigh or left arm deltoid region in participants below 2 years of age, less dominant arm deltoid region in age group 2-45 years
  * Storage Conditions: +2 to +8°C
  Other Names: Vi polysaccharide typhoid vaccine conjugated with Diphtheria toxoid protein
  Arms: Vi-DT Single-dose
Biological: Control Vaccine — * For participant ≥ 1 year one dose of locally licensed Meningococcal conjugate vaccine will be administered
  * For participants 6 months to 1 year one dose of locally licensed Meningococcal conjugate vaccine will be administered during the study and the next dose will be provided after the study unblinding at the completion of 6 months follow up of last subject.
  Other Names: Locally available Meningococcal conjugate vaccine
  Arms: Control

SUMMARY:
This is a multicenter, randomized, observer-blinded, controlled, immune equivalence study of a multi-dose (MD) formulation with 2PE preservative of SK bioscience Vi-DT compared to single dose (SD) formulation without preservative of SK bioscience Vi-DT in participant (6 months - 45 years) including safety population.

The study objectives are as follows:

* Primary objective. Demonstrate the immune equivalence as measured by anti-Vi IgG Geometric Mean Titer (GMT) of multi dose formulation against single dose formulation of Vi-DT (18-45 year age stratum), at 4 weeks after a single dose.
* Secondary objective 1. Demonstrate the immune equivalence as measured by seroconversion rates of anti-Vi IgG antibody titres of multi dose formulation against single dose formulation of Vi-DT vaccine (18-45 year age stratum) at 4 weeks after a single dose.
* Secondary objective 2. Describe safety profile in all age strata combined (age 6 months - 45 years old) and in each age stratum, at 4 weeks after a single dose of SD/MD formulation/control (Meningococcal Conjugate Vaccine).

There are total 5 scheduled visits as follows:

* Visit 1(D-7 to 0): Screening
* Visit 2(D0): Enrollment, vaccination, safety follow-up and blood collection for immunogenicity assessment (only for subjects 18 years old and above)
* Visit 3(D7): Safety follow-up
* Visit 4(D28): Safety follow-up and blood collection for immunogenicity assessment (only for subjects 18 years old and above)
* V5(D168): Safety follow-up

DETAILED DESCRIPTION:
The vaccines will be administered to 1,500 healthy participants of 6 months to 45 years of age and followed up for 24 weeks after the injection for safety. Adult participants (N=500) will be followed up for immunogenicity at 4 weeks and all participants till 24 weeks for safety post single dose of either MD & SD formulations. 300 healthy participants will be given control vaccine (locally available licensed Meningococcal conjugate vaccine) to check the background safety events. The primary objective is to demonstrate the equivalence of immunogenicity as measured by anti-Vi IgG GMT titer at 4 weeks after a single dose of MD/SD formulation in adults. The secondary objective is to demonstrate the equivalence of immunogenicity in terms of seroconversion rates as measured by anti-Vi IgG ELISA antibody titers, at 4 weeks after a single dose of MD/SD formulation in adults. A descriptive evaluation of safety at 4 and 24 weeks post single dose of (SD/MD/Meningococcal vaccine), will be performed. The Vi-DT vaccine from both MD & SD formulations will be administered as a single dose of 25 µg/0.5 mL.

Eligible participants enrolled into the study will be randomized into one of the three study groups within each age stratum of 6 months to less than 2 years, 2 to less than 18 years, and 18 to 45 years. Participants will be observed at the study site for 30 minutes after vaccination for safety assessment. Solicited adverse events will be recorded on a diary card during 7 days after vaccination. Unsolicited adverse events will be recorded during the 4 weeks after vaccination. Serious adverse events will be recorded during the entire study period. With the exception of designated study site personnel responsible for vaccine administration, site investigators, study nurse, and those assessing clinical outcomes, and data analysts will be blinded to vaccine allocation until data base lock for the final analysis.

Blood samples will be collected at baseline prior to vaccination and at 4 weeks post vaccination from adults (18-45 years) for immunogenicity assessment

ELIGIBILITY:
Inclusion Criteria:

1. Healthy participants 6 months to 45 years of age at enrollment
2. Participants/Parent(s)/LAR who have voluntarily given informed consent/assent
3. Participants/Parent(s)/LAR willing to follow the study procedures of the study and available for the entire duration of the study

Exclusion Criteria:

1. Child with a congenital abnormality
2. Participant who has already received meningococcal conjugate vaccine
3. Participants concomitantly enrolled or scheduled to be enrolled in another trial
4. Known history of immune function disorders including immunodeficiency diseases (Known HIV infection or other immune function disorders)
5. Chronic use of systemic steroids (>2 mg/kg/day or >20 mg/day prednisone equivalent for periods exceeding 10 days), cytotoxic or other immunosuppressive drugs
6. Receipt of blood or blood-derived products in the past 3 months
7. Participant with a previously ascertained or suspected disease caused by S. Typhi (confirmed either clinically, serologically or microbiologically)
8. Participant who has had household contact with and/or intimate exposure to an individual with laboratory-confirmed S. Typhi
9. Individual who has previously received a typhoid vaccine
10. Participant who has received other vaccines from 1 month prior to test vaccination or planned to receive any vaccine within 1 month (except a measles containing vaccine as per government vaccination campaign)
11. Known history or allergy to vaccines or other medications
12. History of uncontrolled coagulopathy or blood disorders
13. Any abnormality or chronic disease which in the opinion of the investigator might be detrimental for the safety of the participant and interfere with the assessment of the study objectives
14. Any female participant who is lactating, pregnant* or planning for pregnancy during the course of study period
15. Participants/Parent(s)/LAR planning to move from the study area before the end of study period
16. As per Investigator's medical judgement individual could be excluded from the study in spite of meeting all inclusion/exclusion criteria mentioned above

Ages: 6 Months to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1800 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2020-09-11 (Actual); Study Completion 2021-01-29 (Actual)

PRIMARY OUTCOMES:
Geometric Mean Titers (GMT) of anti-Vi IgG | At 4 weeks (28 days) post vaccination of Vi-DT (MD/SD)
  If the 95% confidence interval of the ratio of GMT estimate of Vi-DT(MD) over GMT of Vi-DT(SD) is located within the bounds of 0.67to 1.5, then Vi-DT (MD) is equivalent to Vi-DT (SD) in terms of GMT of anti-Vi IgG with significance level of 0.05.

SECONDARY OUTCOMES:
Seroconversion rates of anti-Vi IgG ELISA antibody titres | At 4 weeks (28 days) from baseline (Day 0; before vaccination of Vi-DT (MD/SD)
  If the 95% confidence interval of the estimate of difference of seroconversion rate between Vi-DT (MD) and Vi-DT (SD) at 4 weeks (Day 28) is located within the bounds -10% to 10%, then Vi-DT (MD) is equivalent to Vi-DT (SD) in terms of sero-conversion rate, which is defined as 4 fold increase of anti Vi IgG from baseline with significance level of 0.05.

OTHER OUTCOMES:
Safety endpoints by each formulation and overall and within each age stratum | Solicited AEs during the 7 days after vaccination/Unsolicited AEs during 4 weeks (28 days) after vaccination/SAEs during the entire study period
  1. Frequency of local and systemic solicited adverse events during the 7 days after each dose
     * Solicited local reactions at the site of injection: pain, tenderness, erythema/redness, swelling/induration and pruritus
     * Solicited systemic reactions (adapted to each age group): fever, lethargy, irritability, nausea/vomiting, arthralgia, diarrhea, drowsiness, loss of appetite, chills, headache, fatigue, myalgia and persistent crying
  2. Frequency of unsolicited adverse events during 4 weeks (28 days) after vaccination
  3. Frequency of Serious Adverse Events during the entire study period

CONTACTS AND LOCATIONS:
Overall Officials: Josefina C Carlos, MD, Principal Investigator — University of the East-Ramon Magsaysay Memorial Medical Center Inc.
Locations (4):
- Philippines (4):
  - Lingga Health Research Center, Calamba, Laguna
  - Magcase Health Center, San Pablo, Laguna
  - Putatan Research Center, Muntinlupa, National Capital Region
  - University of the Philippines Manila-National Institutes of Health, Manila

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carlos JC, Tadesse BT, Borja-Tabora C, Alberto E, Ylade MC, Sil A, Kim DR, Ahn HS, Yang JS, Lee JY, Kim MS, Park J, Kwon SY, Kim H, Yang SY, Ryu JH, Park H, Shin JH, Lee Y, Kim JH, Mojares ZR, Wartel TA, Sahastrabuddhe S. A Phase 3, Multicenter, Randomized, Controlled Trial to Evaluate Immune Equivalence and Safety of Multidose and Single-dose Formulations of Vi-DT Typhoid Conjugate Vaccine in Healthy Filipino Individuals 6 Months to 45 Years of Age. Lancet Reg Health West Pac. 2022 May 30;24:100484. doi: 10.1016/j.lanwpc.2022.100484. eCollection 2022 Jul. PMID 35664443